CLINICAL TRIAL: NCT02906345
Title: "Analyses on the Effectiveness and Technical Optimization of Therapeutic Plasma Exchange for Patients With Septic Shock, With Special Emphasis on Influencing the Kidney, Liver and Nervous System Through the Extracorporeal Therapy"
Brief Title: TPE in Septic Patients and Influence on Organ Failure
Acronym: TPEMOF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Martin Sauer, MD, PD Dr. med. habil.; MD, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A 2016-0144
Record Dates: First submitted 2016-09-03; First posted 2016-09-20 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Multiple Organ Failure
Keywords: Septic shock; Fresh frozen plasma
MeSH Terms: conditions — Multiple Organ Failure; Shock, Septic | interventions — Plasma Exchange

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (No Intervention): Patients with septic shock, no therapeutic plasma exchange, BMC standard treatment
- TPE-Filtration Group (Active Comparator): Patients with septic shock, therapeutic plasma exchange, plasma separation using a filter (Fresenius MultiFiltrate, Kit 16 MPS P2 dry), BMC standard treatment
  Interventions: Device: Therapeutic Plasma Exchange (TPE)
- TPE-Centrifugation (Active Comparator): Patients with septic shock, therapeutic plasma exchange, plasma separation using a centrifuge (Fresenius COM-TEC, PL1 Erythrozytapherese/Plasmabeutel Set) BMC standard treatment
  Interventions: Device: Therapeutic Plasma Exchange (TPE)

INTERVENTIONS:
Device: Therapeutic Plasma Exchange (TPE) — All treated patients should treated two (minimal) to five times by TPE, depending on the need of norephinephrine for the therapy. For each session 40 ml/kg body weight plasma should be exchange. Fluid resuscitation will be done with fresh frozen plasma.
  Arms: TPE-Centrifugation; TPE-Filtration Group

SUMMARY:
Therapeutic plasma exchange (TPE) should used for patients with septic shock in a controlled, prospective study focusing on the organ functions of the patients.

DETAILED DESCRIPTION:
Therapeutic plasma exchange (TPE) should used for patients with septic shock in a controlled, prospective study.

Investigators will study three groups:

1. untreated control group;
2. TPE group, plasma separation carried out by filtration;
3. TPE group, plasma separation carried out by centrifugation.

All treated patients should treated two (minimal) to five times by TPE, depending on the need of norephinephrine for the therapy. For each session 40 ml/kg body weight plasma should be exchange. Fluid resuscitation will be done with fresh frozen plasma. The study will focusing on the organ functions of the patients, especially liver-, kidney- and nervous function and also displayed in the SOFA score on study days 3 and 7.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock, beginning of shock < 24 hours

Exclusion Criteria:

* Participation in an another clinical trial within the last 30 days
* Participation in this study at an earlier date
* Simultaneous participation in another clinical trial
* Pregnancy
* Unpredictable Bleeding (over 2 erythrocyte concentrates daily)
* Polyneuropathy (known before the beginning of sepsis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-04 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
SOFA score ≥ 2 Punkte | day 3
  SOFA: Sepsis-related Organ Failure Assessment score
SOFA score ≥ 2 Punkte | day 7
  SOFA: Sepsis-related Organ Failure Assessment score

SECONDARY OUTCOMES:
28-day survival | day 28
  Observation time 28 days
Hospital survival | 1 year
  Leave the patients the hospital?

OTHER OUTCOMES:
number of thrombocytes (DIC) | days 1-7, 14, 21, 28
  values of thrombocytes, screening for DIC
Haptoglobulin values | days 1-7, 14, 21, 28
  values haptoglobulin, screening for hemolysis

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Units PIT 1+2, University Hospital Rostock, Rostock, Germany

IPD SHARING:
Plan to Share IPD: No
No.